CLINICAL TRIAL: NCT03151265
Title: A Prospective Open Label Pilot Study Investigating the Impact of ThermaCare on Flexibility, Muscle Relaxation & Low Back Pain in Two Different Populations
Brief Title: A Prospective Pilot Study Investigating the Impact of ThermaCare on Flexibility, Muscle Relaxation & Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: dorsaVi Ltd (Industry)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017THERMA
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-04

CONDITIONS: Low Back Pain
Keywords: Functional Outcome Measures; Wearable Sensors; ViMove; Low Back Pain; Range of Movement; Muscle Activity; ThermaCare
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: The two study groups (LBP group vs. Active in spot group), will receive the same intervention in the same order (i.e. Baseline day with no intervention, then intervention day with ThermaCare intervention).
Masking Description: This study is open label, meaning that no masking occurs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Low Back Pain Group (Experimental): Low Back Pain (LBP) group will be assessed on two consecutive days. The first day will have no ThermaCare intervention applied, and is for a Baseline assessment of flexibility, muscle relaxation and low back pain.
  The second day will have the ThermaCare Low Back Heat Wrap intervention applied, and will have the same assessments as the Baseline day.
  Interventions: Device: ThermaCare Low Back Heat Wrap
- Active in Sport Group (Experimental): Sport group will be assessed on two consecutive days. The first day will have no ThermaCare intervention applied, and is for a baseline assessment of flexibility, muscle relaxation and low back pain.
  The second day will have the ThermaCare Low Back Heat Wrap intervention applied, and will have the same assessments as the Baseline day.
  Interventions: Device: ThermaCare Low Back Heat Wrap

INTERVENTIONS:
Device: ThermaCare Low Back Heat Wrap — The ThermaCare Low Back Heat Wrap, is a continuous, low-level, direct heat therapy. It comes in the form of a heat-pack that is strapped to the low back. Heat is provided for approximately 8-hours.

SUMMARY:
The objective of this Investigator Initiated study is to evaluate the effectiveness of ThermaCare HeatWraps in improving flexibility and low back muscle relaxation, and in participants experiencing pain, reducing pain during movement. This study is an intervention trial on two discrete subject samples; (1) people with recent back pain, and (2) people who regularly play sport. ViMove wearable sensors provide precise objective measurements of low back muscle activity and movement in real time and can capture a patient's reporting of pain during movement. Outcomes will be assessed through standard ViMove protocols in conjunction with multiple validated measures of pain, perception of change, and function.

DETAILED DESCRIPTION:
This investigator-initiated study will utilize a prospective open-label study design to evaluate the effectiveness of ThermaCare HeatWraps in improving flexibility and low back muscle relaxation, and in participants experiencing pain, reducing pain during movement. Two discrete subject samples will be enrolled; (1) people with recent back pain, and (2) people who regularly play sport. Both samples will be enrolled using respective criteria.

Following enrollment, both subject groups will have a "start interview" on their allocated baseline assessment day (Day 1). This will include fitting of the ViMove movement and EMG sensors, as well as a live "pain on movement" assessment. This session will take approximately 20-30 minutes. Whilst wearing the ViMove sensors, subjects will then leave the clinic and conduct normal daily activities for a pre-determined monitoring period. No ThermaCare HeatWraps are worn on Day 1. This allows a baseline assessment and allows any placebo effects from the sensors to be discounted. At the end of the monitoring session, subjects will return to the clinic to have an "end-of-day" interview. Clinicians will administer the Oswestry Disability Index (ODI), the Visual Analogue Scale for Pain (VAS Pain), and the Patient Global Impression of Change scale (PGIC). ViMove movement sensors will then be removed, and the subject will be reimbursed for that day.

The intervention day (Day 2) will have the same procedure as Day 1 (baseline), with the only difference being the additional application of ThermaCare HeatWraps during the "start interview". Subjects will continue to wear the HeatWrap and ViMove sensors during the 8-hour daily activity monitoring period, with the wrap and sensors being removed during the end-of-day interview. The subject will then be reimbursed for Day 2.

ELIGIBILITY:
Inclusion criteria for recent low back pain patients (Group 1):

1. Adults between the age of 21-54 inclusive, male and female.
2. Low back pain is the primary source of pain over the last 3 weeks.
3. Have experienced and received treatment for muscle related low back pain with an average score of at least 3/10 on a 10-point Numeric Rating scale over the past 3 weeks.
4. Must be able to communicate fluently in English.
5. Must provide written informed consent.
6. Must agree to confidentiality.

Inclusion criteria for people who are active in sports (Group 2):

1. Adults between the age of 21-54 inclusive, male and female.
2. Participate in 30 min of moderate to high intensity exercise 3 times per week. As defined by Borg Rating of Perceived Exertion scale.
3. Must be able to communicate fluently in English.
4. Must provide written informed consent.
5. Must agree to confidentiality.

Exclusion Criteria (applies to both Groups):

1. The subject is pregnant.
2. The subject has a severe hearing impairment.
3. The subject is cognitively impaired.
4. Known allergic skin reaction to tapes and plasters.
5. Co-morbidities of neoplasm, infection, fracture, inflammatory or metabolic disorder that has potential to affect the lumbo-pelvic region.
6. Person who is currently enrolled in another investigational drug or device study.

Ages: 21 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ronchi, PhD, Principal Investigator — dorsaVi Ltd
Locations (3):
- Australia (3):
  - Clifton Hill Physiotherapy, Clifton Hill, Victoria
  - Peak MSK Physiotherapy, Hampton, Victoria
  - Hoppers Physio, Hoppers Crossing, Victoria

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Back Pain Group: Low Back Pain (LBP) group will be assessed on two consecutive days. The first day will have no ThermaCare intervention applied, and is for a Baseline assessment of flexibility, muscle relaxation and low back pain.
  The second day will have the ThermaCare Low Back Heat Wrap intervention applied, and will have the same assessments as the Baseline day.
  ThermaCare Low Back Heat Wrap: The ThermaCare Low Back Heat Wrap, is a continuous, low-level, direct heat therapy. It comes in the form of a heat-pack that is strapped to the low back. Heat is provided for approximately 8-hours.
- Active in Sport Group: Sport group will be assessed on two consecutive days. The first day will have no ThermaCare intervention applied, and is for a baseline assessment of flexibility and muscle relaxation.
  The second day will have the ThermaCare Low Back Heat Wrap intervention applied, and will have the same assessments as the Baseline day.
  ThermaCare Low Back Heat Wrap: The ThermaCare Low Back Heat Wrap, is a continuous, low-level, direct heat therapy. It comes in the form of a heat-pack that is strapped to the low back. Heat is provided for approximately 8-hours.
Period: Overall Study
Arm/Group | Low Back Pain Group | Active in Sport Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active in Sport Group: Sport group will be assessed on two consecutive days. The first day will have no ThermaCare intervention applied, and is for a baseline assessment of flexibility, muscle relaxation and low back pain.
  The second day will have the ThermaCare Low Back Heat Wrap intervention applied, and will have the same assessments as the Baseline day.
  ThermaCare Low Back Heat Wrap: The ThermaCare Low Back Heat Wrap, is a continuous, low-level, direct heat therapy. It comes in the form of a heat-pack that is strapped to the low back. Heat is provided for approximately 8-hours.
- Total: Total of all reporting groups
Arm/Group | Low Back Pain Group | Active in Sport Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 4 | 9 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Movement Data Over Time
Description: Collection of movement data from all participants. The results listed here depict the average change in Trunk Range of Motion (ROM) between day 1 and day 2 PM sessions
Time Frame: Change from Baseline movement data after 1 consecutive day.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Low Back Pain Group | Active in Sport Group
Number analyzed (Participants) | 20 | 20
Degrees | 2.74 (6.17) | 1.1 (6.9)

2. Primary Outcome: Change in Erector Spinae Muscle Activity Over Time
Description: Collection of erector spinae muscle activity data from all participants. The results provided depict the mean muscle-activity difference between the day 1 and day 2 PM sessions.
  Surface Electromyography (sEMG) sensors are adhered utilizing a height-specific sensor placement template. Placement is parallel with the L3 vertebrae.
  Evaluated in the form of the flexion-relaxation response. When performing a forward flexion movement, muscle activation occurs at the commencement of the movement (when bending down;concentric), as well as during the return to the upright position (eccentric). At maximum flexion, minimal muscle activation is expected (i.e. muscle relaxation). However, in subjects with Low-back pain, muscle relaxation is often absent.
  As such, the following formula is used to evaluate the flexion-relaxation response.
  Sum of sEMG activity at maximum flexion divided by the summed sEMG activity of both concentric and eccentric muscle activation.
Time Frame: Change from Baseline Erector spinae muscle activity data after 1 consecutive day.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Low Back Pain Group | Active in Sport Group
Number analyzed (Participants) | 20 | 20
Ratio | -.13 (.28) | -.019 (.45)

3. Secondary Outcome: A Change Over Time in Range of Motion in Any One Plane of Movement Compared to Pre-intervention Range of Motion.
Description: Maximal range of low back movement in sagittal,axial and coronal planes. Results depict the change in Pelvis ROM in the sagittal plane.
Time Frame: Change from Baseline after 1 consecutive day.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Low Back Pain Group | Active in Sport Group
Number analyzed (Participants) | 20 | 20
Degrees | 2.05 (6.6) | 3.11 (7.8)

4. Secondary Outcome: In Group 1 (LBP Patients), a Change in Maximum Pain During Movement Score, for Any One Plane of Movement.
Description: Pain Score out of 10 as rated on the ViMove scale during movement assessment. Score from 0-10 where 10 indicates maximum pain, and 0 indicates no pain. The results depicted indicate the change in pain scores between baseline and post-intervention
Time Frame: Change from Baseline after 1 consecutive day.
Population: Pain scores were not captured for the sports group as 'no pain' is a selection criterion for this group.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Low Back Pain Group | Active in Sport Group
Number analyzed (Participants) | 20 | 0
score on a scale | .3 (.58) |

5. Secondary Outcome: A Change in Muscle Activity From Baseline in Subjects Where Abnormal EMG Activity During Baseline is Detected.
Description: Surface EMG measurement of erector spinae muscle activity at L3 vertebra level
Time Frame: Change from Baseline after 1 consecutive day.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Low Back Pain Group | Active in Sport Group
Number analyzed (Participants) | 20 | 20
Ratio | -.13 (.28) | -.019 (.45)

6. Secondary Outcome: Change in Pain From Baseline
Description: Pain Score out of 10 as measured on a Numeric Rating scale (NRS)
  Score from 0-10 where 10 indicates maximum pain, and 0 indicates no pain.
  The results depicted indicate the change in NRS scores between baseline and post-intervention
Time Frame: Change from Baseline after 1 consecutive day.
Population: Pain scores were not captured for the sports group as 'no pain' is a selection criterion for this group.
Measure: Mean (Standard Error); unit: scale on a scale
Arm/Group | Low Back Pain Group | Active in Sport Group
Number analyzed (Participants) | 20 | 0
scale on a scale | -.1 (.71) |

7. Secondary Outcome: Observation of Self-reported Changes in Functional Status Pre- and Post- ThermaCare Application as Measured by the Oswestry Disability Index (ODI) if Subjects Scored >3 on the NRS
Description: Measurement of disability related to low back pain. Contains 10 sections, each of which can be from from 0-5 for a maximum score of 50.
  50 indicates maximum possible disability (bed-bound - or are exaggerating their symptoms).
  The results depicted indicate the change in NRS scores between baseline and post-intervention
Time Frame: Change from Baseline after 1 consecutive day.
Population: ODI scores were not captured for the sports group as 'no pain/disability' is a selection criterion for this group.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Low Back Pain Group | Active in Sport Group
Number analyzed (Participants) | 20 | 0
score on a scale | .70 (2.29) |

8. Secondary Outcome: Impression of Change From Subjects Post Intervention and/or Assessment Period Using the Patient Global Impression of Change Scale (PGIC).
Description: Measurement of perceived change in Low back pain. Score from a scale of 1-7. 1 indicates no change (or condition has worsened), 7 indicates a considerable improvement.
  The results depicted indicate the change in PGIC scores between Day 1 and Day 2 (intervention)
Time Frame: Change from Baseline after 1 consecutive day.
Population: PGIC data were not collected for the Active in Sport Group, as subjects in this group were selected on the basis that they had no pain. As such, they would not have had an applicable impression of change related to pain.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Low Back Pain Group | Active in Sport Group
Number analyzed (Participants) | 20 | 0
score on a scale | 2.7 (.45) |

9. Secondary Outcome: Observation of Self-reported Changes in Functional Status Pre- and Post- ThermaCare Application as Measured by the Roland Morris Disability Questionnaire (RMDQ) if Subjects Scored >3 on the NRS
Description: Measurement of disability related to low back pain. A checklist of 24 items. A score of 24 indicates maximum disability.
Time Frame: Change from Baseline after 1 consecutive day.
Population: RMDQ scores were not captured for the sports group as 'no pain/disability' is a selection criterion for this group.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Low Back Pain Group | Active in Sport Group
Number analyzed (Participants) | 20 | 0
score on a scale | .20 (2.00) |

ADVERSE EVENTS:
Time Frame: From the 10th July 2017 to the 23rd December 2017. This is from the first assessment date, to two days after the final assessment date.
Arm/Group | Low Back Pain Group | Active in Sport Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-05-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT03151265/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-05-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT03151265/Prot_SAP_001.pdf